CLINICAL TRIAL: NCT00970658
Title: Clinical Multicenter Study, Randomized, Open, to Evaluate the Efficacy and Safety of Salonsip Compared to Sabiá Plaster Relief of the Signs and Symptoms in Patients With Contusions, Sprains, Injuries and Muscular Injuries With Less Than 24 Hours Early or Holders of Myalgia, Pain and Tendonitis in Regions Miofasciais Articulated.
Brief Title: Efficacy and Safety of Salonsip Compared to Sabiá Plaster
Acronym: SAL-SIP-03/09
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hisamitsu Farmaceutica do Brasil Ltda (Industry)
Responsible Party: Emília Wakebe, Hisamitsu Farmacêutica do Brasil Ltda.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAL-SIP-03/09
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Contusions; Sprains; Myalgia; Pain; Tendonitis
Keywords: Plaster; injuries; regions miofasciais articulated; Reducing signs, symptoms
MeSH Terms: conditions — Contusions; Sprains and Strains; Myalgia; Pain; Tendinopathy; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Salonsip (Experimental): The plaster should be applied at the site of injury, which must be clean and dry and changed every 8 hours for a period of 48 hours of treatment (2 days).
  Interventions: Drug: Salonsip plaster
- Sabiá (Active Comparator): The plaster should be applied at the site of injury, which must be clean and dry and changed every 8 hours for a period of 48 hours of treatment (2 days).
  Interventions: Drug: Sabia plaster

INTERVENTIONS:
Drug: Salonsip plaster — The plaster should be applied at the site of injury, which must be clean and dry and changed every 8 hours for a period of 48 hours of treatment (2 days).
  Arms: Salonsip
Drug: Sabia plaster — The plaster should be applied at the site of injury, which must be clean and dry and changed every 8 hours for a period of 48 hours of treatment (2 days).
  Arms: Sabiá

SUMMARY:
The purpose of this study is to evaluate the efficacy in reducing signs and symptoms in patients with contusions, sprains, muscular injuries and injuries with less than 24 hours early or holders of myalgia, pain and tendonitis in regions miofasciais articulated with Salonsip compared to Sabiá plaster.

It is clinical, open, multicenter, randomized, prospective and comparative, with patients entering at random.

Patients will be included in sufficient quantity to achieve the minimum number of 70 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, of any race, aged 12 years;
* Ability to read, understand and sign the Consent Form, in the case of children under age monitoring and consent of the person responsible;
* Clinical diagnosis of bruises, sprains, trauma, muscle damage occurring in times less than 24 hours or myalgia, pain miofasciais or tendonitis.
* Patients able to understand and maintain the clinical protocol

Exclusion Criteria:

* Known hypersensitivity to components of the formulas of both the product and the comparative test.
* Known hypersensitivity to paracetamol.
* Location of the lesion with skin wound or irritated.
* Hepatic or renal diseases known.
* Pregnant or breastfeeding.
* Patients who require surgery or immobilization rigid;
* Patients with fractures or rupture of the ligaments.
* Patients in use of anticoagulants.
* Patients with severe concomitant systemic diseases such as cancer, diabetes, congenital or acquired heart disease, hematological diseases, convulsive disorders, autoimmune diseases, renal failure, infections, hormonal disorders and pulmonary disorders.
* History of alcoholism or use of illicit drugs;
* Use of non-steroidal anti-inflammatory drugs, corticosteroids or venoterápicos, topics or any other form of administration.
* Conditions which in the opinion of the investigator makes the patient unsuitable to participate in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-01 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Likert Scales and Visual Analogue Scales | two days

SECONDARY OUTCOMES:
Safety evaluation by adverse events relate. | two days